CLINICAL TRIAL: NCT02695732
Title: Primary Prophylaxis of High-risk Esophageal Gastric Variceal Bleeding Comparing Carvedilol and Endoscopic Therapy: A Multicenter Randomized Controlled Trial
Brief Title: The Effect of Carvedilol VS Endoscopic Therapy in Primary Prophylaxis of High-risk Esophageal Gastric Variceal Bleeding
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai Public Health Clinical Center (Other Government); ShuGuang Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Gongli Hospital, School of Medicine, The Second Military Medical University (Unknown); Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, Shiyao Chen, Director of department of Gastroenterology, Zhongshan Hospital, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSY-LC02-2016
Record Dates: First submitted 2016-02-25; First posted 2016-03-01 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Liver Cirrhosis; Esophageal and Gastric Varices
Keywords: Esophageal and Gastric Varices; Primary Prophylaxis; Carvedilol; Endoscopy
MeSH Terms: conditions — Liver Cirrhosis; Esophageal and Gastric Varices | interventions — Carvedilol; Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carvedilol (Experimental): Carvedilol，6.25mg-12.5mg/d,oral,6-36 months
  Interventions: Drug: Carvedilol
- endoscopy (Active Comparator): endoscopy，every 4 weeks until eradication of varices
  Interventions: Device: endoscopy

INTERVENTIONS:
Drug: Carvedilol — Carvedilol is started at a dose of 6.25 mg/d, and titrated to a maximum dose of 12.5 mg/d.Doses are increased every 7 days until ABPsys is not less than 95 mm Hg and HR is not less than 55 bpm.
  Other Names: JinLuo; LvDao
  Arms: Carvedilol
Device: endoscopy — Patients receiving endoscopic therapy (either endoscopic ligation or cyanoacrylate injection) every 4 weeks until eradication of varices.
  Arms: endoscopy

SUMMARY:
To compare the efficacy and safety of Carvedilol and endoscopic therapy in Primary Prophylaxis of High-risk Esophageal Gastric Variceal Bleeding.

DETAILED DESCRIPTION:
The study is a randomized controlled trial. Patients randomly enter into two treatment groups: 1)the Carvedilol group and 2)the endoscopy group. Treatment allocation is by block randomization, with an two-to-one ratio for Carvedilol and endoscopy. The results are concealed in opaque envelopes. The dose of Carvedilol is titrated according to systolic arterial blood pressure (ABPsys) and heart rate (HR). Doses are increased every 7 days until ABPsys is not less than 95 mm Hg and HR is not less than 55 bpm. Carvedilol is started at a dose of 6.25 mg/d, and titrated to a maximum dose of 12.5 mg/d. Patients receiving endoscopic therapy every 4 weeks until eradication of varices. Patients will come for clinic visit every 6 months, receiving laboratory tests and endoscopic examinations, and events of primary and secondary outcomes will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* the presence of severe esophageal and gastric varices at upper gastrointestinal endoscopy without a previous haemorrhage
* a diagnosis of liver cirrhosis based on histology, clinical or imaging manifestation

Exclusion Criteria:

* age greater than 80 years old or younger than 18 years old
* non-cirrhotic portal hypertension
* contraindications to NSBB including bronchospasm, severe bradycardia, severe heart failure, acute pulmonary edema, atrioventricular block and so on
* ABPsys less than 95 mmHg or HR less than 50 bpm
* prior treatment for prevention of bleeding from EGV
* presence of spontaneous bacterial peritonitis or other severe infections
* presence of hepatorenal syndrome
* uncontrolled hepatic encephalopathy
* presence of refractory ascites
* pregnancy
* presence of portosystemic shunt or portal cavernous transformation
* refusal to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 792 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Bleeding rate | through study completion，an average of 18 months
  The investigators observe the variceal bleeding events during the study

SECONDARY OUTCOMES:
Mortality rate | through study completion，an average of 18 months
  The investigators observe the mortality events during the study due to variceal bleeding, hepatic encephalopathy, liver failure, hepatic cellular carcinoma, hepatic-renal syndrome and spontaneous bacterial peritonitis.
Adverse events | through study completion，an average of 18 months
  The investigators observe any severe adverse events caused by drug or endoscopic treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Shiyao Chen, Professor, Study Director — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan Hospital, Shanghai, China